CLINICAL TRIAL: NCT06552975
Title: Transcriptome-based Diagnostic Biomarker for Acute Febrile Illness: a Cross-sectional Observational Study
Brief Title: Clinical Study of Transcriptome-based Diagnostic Biomarker for Acute Febrile Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202008-058
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2023-11

CONDITIONS: Acute Febrile Illness
Keywords: Bacterial infection; Viral infection; noninfectious disease
MeSH Terms: conditions — Bacterial Infections; Virus Diseases; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 2-3ml of peripheral blood samples collected by each patient were divided into two parts, one part was added with trizol for subsequent RT-PCR, and the other part was used for separating serum and detecting serum biomarker.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bacterial infection: Individuals with acute fever whose positive bacteria isolated from sterile or non-sterile sites have pathological characteristics.
  Interventions: Other: Infection
- Viral infection: Individuals with acute fever whose viral nucleic acid test and/or serological positive compatible with acute syndrome#(e.g. serology, PCR).
  Interventions: Other: Infection
- non-infectious group: Individuals with acute fever whose have negative findings in cultures and PCR; negative image modality findings suspected for infection; confirmed or highly likely other diagnosis; improvement without antibiotics.

INTERVENTIONS:
Other: Infection — Pathogens such as bacteria and viruses invade the human body, grow, and proliferation, triggering an immune response.
  Groups: Bacterial infection; Viral infection

SUMMARY:
Acute febrile illness is the main cause of outpatient visits，and bacterial and viral infections remains the most common cause. The diagnosis of infection is still based on symptoms and traditional techniques, resulting in overuse of antibacterial drugs or delay in treatment. The signature of host transcripts has a potential to reveal different modes of host-pathogen interaction and may serve as a biomarker for infection discrimination. Of note, transcriptome-microarray and RNA-seq methods need sophisticated techniques and expertise interpretation, hampering the universal implement of these platforms in low-tier hospitals and under- resourced countries. This study explores transcriptome-based diagnostic biomarker for acute febrile illness , hoping to achieve rapid, accurate and cost-effective distinction between bacterial and viral infection.

DETAILED DESCRIPTION:
Acute fever is a common medical emergency worldwide, most often caused by bacterial or viral infections. Early and rapid differential diagnosis of infectious diseases is crucial for improving patient outcomes. While pathogen detection remains the gold standard for diagnosing infections, methods like culture are time-consuming and often lack sensitivity. Additionally, the presence of normal colonizing microorganisms, such as bacteria and viruses in the human body, can lead to false positives in pathogen detection. These limitations often compel physicians to rely on empirical antibacterial therapy based on clinical symptoms, inadvertently contributing to antibiotic overuse and the growing problem of bacterial resistance.

Furthermore, the misuse of antibacterial drugs in patients with non-bacterial infections can lead to complications such as secondary infections with Clostridium difficile, liver dysfunction, kidney damage, cytopenia, and alterations in the body's microbiota. Diagnostic markers based on host inflammatory responses offer an alternative approach to infection diagnosis. However, protein biomarkers like procalcitonin, though widely used in clinical settings, are far from ideal for accurately diagnosing bacterial infections, as they are prone to false positives and negatives.

A promising direction is the analysis of host-pathogen interactions at the transcriptome level, particularly the differential gene expression of the host in response to various pathogens. This area of research has gained significant attention recently. Transcriptomic markers derived from patients' peripheral blood have been successfully utilized in diagnosing and studying the pathogenesis of various infectious diseases.

Despite these advances, studies relying on RNA sequencing or transcriptome chip technology require specialized equipment and bioinformatics expertise, making them expensive and challenging to implement in routine clinical practice. Additionally, the results from transcriptome analysis are not easily validated by reverse transcription polymerase chain reaction(RT-PCR), the "gold standard" for RNA quantification. Therefore, to make transcriptome-based diagnostic markers more clinically applicable, there is a need for real-time technologies, such as PCR, to enhance the accuracy of infection diagnosis and reduce the misuse of antibacterial drugs. Currently, research in this area remains limited.

ELIGIBILITY:
Inclusion Criteria:

* 1. axillary temperature ≥38°C; 2. duration of fever shorter than 14 days; 3. subjects who are fully informed and agree to participate in this study.

Exclusion Criteria:

* 1.having comorbidities that may affect host gene expression, such as advanced malignancy, autoimmune diseases，immunodeficiency, or taking immune suppressors; 2.pregnancy; 3. mixed infection (viral combined with bacterial infection, autoimmune disease combined with bacterial infection); 4.incomplete clinical information; 5. For safety reasons or the interests of patients, clinicians believe that patients should not participate in any situation in this study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who have an axillary temperature of 38°C or higher, with a fever duration of less than 14 days.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
AUC for distinguishing bacterial infection from viral infection | Through study completion, an average of 2 years
  The AUC of the transcript biomarkers for distinguishing bacterial infection from viral infection reflects the diagnostic accuracy of the transcript biomarkers.

SECONDARY OUTCOMES:
AUC for distinguishing infectious disease from noninfectious disease | Through study completion, an average of 2 years
  The AUC of the transcript biomarkers for distinguishing infectious disease from noninfectious disease reflects the diagnostic accuracy of the transcript biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
It may require further evaluation of data privacy and ethical considerations to ensure that participants' privacy is not compromised by data sharing.